CLINICAL TRIAL: NCT02183623
Title: The Effect of Multiple Oral Doses of BI 1356 BS as Tablets Once Daily for Six Days on the Pharmacokinetics, Safety and Tolerability of Multiple Oral Doses of 40 mg Simvastatin Given Once Daily for 20 Days and on the Pharmacokinetics of Its Metabolite Simvastatin Acid. An Open-label Study in Healthy Male Volunteers.
Brief Title: The Effect of Multiple Oral Doses of BI 1356 BS on Pharmacokinetics, Safety and Tolerability of Multiple Oral Doses of Simvastatin and on the Pharmacokinetics of Its Metabolite Simvastatin Acid in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.9
Record Dates: First submitted 2014-07-07; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Simvastatin; Linagliptin

ARMS (1):
- BI 1356 BS and Simvastatin (Experimental)
  Interventions: Drug: Simvastatin; Drug: 10 mg BI 1356 BS

INTERVENTIONS:
Drug: Simvastatin
Drug: 10 mg BI 1356 BS

SUMMARY:
Investigation of the multiple dose pharmacokinetics, safety and tolerability of simvastatin and simvastatin acid with and without concomitant administration of BI 1356 BS

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the following criteria: No findings deviating from normal and of clinical relevance as well as no evidence of a clinically relevant concomitant disease based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), clinical laboratory tests
* Age ≥21 and Age ≤65 years
* BMI ≥18.5 and BMI ≤29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or-neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs, including herbal products, which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of study centre
* Not willing to use adequate contraception (condom use plus another form of contraception e.g. spermicide, oral contraceptive taken by female partner, sterilisation, intrauterine device) during the whole study period from the time of the first intake of study drug until one month after the last intake

Ages: 21 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-09; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration-time curve of simvastatin in plasma at steady state over a uniform dosing interval τ) | up to 600 hours after first administration
Cmax,ss (maximum measured concentration of simvastatin in plasma at steady state over a uniform dosing interval τ) | up to 600 hours after first administration

SECONDARY OUTCOMES:
Tmax,ss (time from last dosing to maximum concentration of the analyte in plasma at steady state) | up to 600 hours after first administration
Cmin,ss (minimum concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | up to 600 hours after first administration
Cpre,N (predose concentration of the analyte in plasma at steady state immediately before administration of the next dose N) | up to 600 hours after first administration
λz,ss (terminal rate constant in plasma at steady state) | up to 600 hours after first administration
t1/2,ss (terminal half-life of the analyte in plasma at steady state) | up to 600 hours after first administration
MRTpo,ss (mean residence time of the analyte in the body at steady state after oral administration) | up to 600 hours after first administration
CL/F,ss (apparent clearance of the analyte in the plasma after extravascular administration at steady state) | up to 600 hours after first administration
Vz/F,ss (apparent volume of distribution during the terminal phase λz at steady state following extravascular administration) | up to 600 hours after first administration
AUCτ,ss (area under the concentration-time curve of simvastatin acid and BI 1356 BS in plasma at steady state over a uniform dosing interval τ) | up to 600 hours after first administration
Cmax,ss (maximum measured concentration of simvastatin acid and BI 1356 BS in plasma at steady state over a uniform dosing interval τ) | up to 600 hours after first administration
Number of patients with adverse events | up to day 30
Clinically relevant changes in clinical laboratory values | up to day 30
Assessment of tolerability by investigator on a 4-point scale | up to day 30